CLINICAL TRIAL: NCT04369482
Title: Posterior Capsule Opafication of Different Hydrophobic Acrylic Intraocular Lenses: Vivinex iSert P261 vs.Clareon IOL
Acronym: Clarinex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Clinical Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Clarinex 1560/2014
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Age Related Cataracts

STUDY DESIGN:
Intervention Model Description: The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. Cataract surgery with precedent bilateral randomized IOL implantation will be performed in subjects who have signed an informed consent form. Postoperative examinations will be implemented in accordance with the approved Investigational Plan on subjects and includes: visual acuity, slitlamp examination, fibrosis, posterior capsule opacification (PCO) score and YAG capsulotomy rate.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcon Clareon (Active Comparator): Implantation of an intraocular lens Alcon Clareon
  Interventions: Device: Hoya Vivinex
- Hoya Vivinex (Active Comparator): Implantation of an intraocular lens Hoya Vivinex
  Interventions: Device: Alcon Clareon

INTERVENTIONS:
Device: Alcon Clareon — Implantation of an intraocular lens Alcon Clareon
  Arms: Hoya Vivinex
Device: Hoya Vivinex — Implantation of an intraocular lens Hoya Vivinex
  Arms: Alcon Clareon

SUMMARY:
On the day of surgery, the first eye to be operated is randomised to receive a Vivinex , HOYA Surgical Optics GmbH or an Clareon, Alcon, Fort Worth, Texas. The second eye to be operated receives the other IOL type.

A complete biomicroscopic examination, visual acuity testing using autorefractometer, contrast sensitivity testing, and standardised retroillumination photography for PCO evaluation, will be performed 6 month (30-60 days), 1.5 years (± 3 months) and 3 (± 3 months) years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract for which phacoemulsification extraction and posterior IOL implantation has planned
* Age 50 and older
* Visual potential in both eyes of 20/30 or better as determined by investigators estimation
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Preceding intraocular surgery or ocular trauma
* Relevant other ophthalmic diseases (such as pseudoexfoliation, glaucoma, uveitis, retinal degenerations, etc.)
* Laser treatment
* Uncontrolled systemic or ocular disease
* Infectious disease
* Pregnancy/Nursing

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
PCO score | 3 years
  subjectively and objectively graded: 0-10 (0= no PCO, 10= maximum PCO)

SECONDARY OUTCOMES:
Visual Acuity | 3 years
  UCDVA(uncorrected distance visual acuity), BCDVA (best corrected distance visual acuity)
Fibrosis | 3 years
  grade of fibrosis assessed subjectively at the slitlamp (grade 0=no fibrosis, grade 3=maximum fibrosis)
Subjective glistening score | 3 years
  neg, <10, 10-20, 20-30, 30-40, >40 uniform or localized
YAG capsulotomy rate | 3 years
  described subjectively at the slitlamp: was a YAG capsulotomy performed yes/no

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna Allgemeines Krankenhaus, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leydolt C, Schartmuller D, Schwarzenbacher L, Prenner V, Danzinger V, Lisy M, Abela-Formanek C, Menapace R. Posterior capsule opacification with two similar-design hydrophobic acrylic intraocular lenses: 3-year results of a randomized controlled trial. J Cataract Refract Surg. 2024 Dec 1;50(12):1242-1246. doi: 10.1097/j.jcrs.0000000000001539. PMID 39137100